CLINICAL TRIAL: NCT00279669
Title: Ultrasound to Detect Evidence for Retinal Detachment in Retinopathy of Prematurity
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Columbia University (Other)
Responsible Party: Dan H. Kauffmann-Jokl, MD, Columbia Presbyterian Medical Center
Other Study IDs: ROP
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of Prematurity; Ultrasound; Eye
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ultrasound examination — contact ultrasound examination
  Other Names: Quantel Cinescan

SUMMARY:
Premature infants stand a risk of danger to the layer of the eye that creates sight that, if untreated, can cause severe vision problems, leading to blindness in some cases. This research study will use ultrasound to examine the eye for retinal changes of prematurity.

DETAILED DESCRIPTION:
Retinopathy of prematurity requires the early detection of retinopathy in neonates with a gestational age of < 28 weeks and a birth weight <1500 g. These evaluations require pupillary dilation, diagnostic expertise, consume much time and expense and are not without morbidity.

B-scan ultrasonography using a hand-held probe is part of the current ophthalmologist's armamentarium, providing a non-invasive view of the eye and avoiding the morbidity associated with mydriatic drops used for pupillary dilation.

We will use a simple water bath enclosure for a standard 20 MHz probe currently in general ophthalmic use to determine whether this simple technique might supplant indirect ophthalmoscopy as a screening technique. We will compare, using masked observers, the clinical findings of indirect ophthalmoscopy of neonatal infants with ultrasonic findings to determine if a correlation in the stages of retinopathy of prematurity (ROP) between the two techniques existed.

ELIGIBILITY:
Inclusion Criteria:

premature birth

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premature babies with Retinopathy of Prematurity
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2004-12; Primary Completion 2010-04-30 (Actual); Study Completion 2010-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan H Kauffmann-Jokl, MD, Principal Investigator — Columbia University; Ronald H Silverman, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Columbia Presbyterian Medical Center, New York, New York, United States

REFERENCES:
- [Result] Jokl DH, Silverman RH, Springer AD, Towers H, Kane S, Lopez R, Chiang MF, Lloyd HO, Barbazetto I, Horowitz R, Vidne O. Comparison of ultrasonic and ophthalmoscopic evaluation of retinopathy of prematurity. J Pediatr Ophthalmol Strabismus. 2004 Nov-Dec;41(6):345-50. doi: 10.3928/01913913-20041101-06. PMID 15609519
- [Result] Jokl DH, Silverman RH, Nemerofiky SL, Kane SA, Chiang MF, Lopez R, Lee G. Is there a role for high-frequency ultrasonography in clinical staging of retinopathy of prematurity? J Pediatr Ophthalmol Strabismus. 2006 Jan-Feb;43(1):31-5. doi: 10.3928/01913913-20060101-04. PMID 16491723
- [Result] D. H. Kauffmann Jokl, R. H. Silverman, IV, S. Kane, R. Lopez, M. F. Chiang, and S. L. Nemerofsky. Cribside Ultrasonography for the Early Detection of Rapidly Progressive Zone 1 ROP Retinal Detachment: Implications for Early Surgical Intervention. Invest. Ophthalmol. Vis. Sci. 2007 48: E-Abstract 3094.